CLINICAL TRIAL: NCT07142590
Title: Iron Balance in Humans Living at High Altitude: Defining Requirements and Optimal Biomarker Thresholds Using a Novel Body Iron Labelling Technique Based on Stable Iron Isotopes.
Brief Title: Determination of Iron Absorption and Losses in People Living at High Altitude to Investigate the Requirements in This Population Group Using a Newly Developed Technique
Acronym: ARIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diego Moretti (Other)
Collaborators: Swiss Federal Institute of Technology (Other); University of Lausanne (Other)
Responsible Party: Sponsor-Investigator, Diego Moretti, Prof. Dr. Diego Moretti, Swiss Distance University of Applied Sciences
Organization: Swiss Distance University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Iron_ARIA_2024
Record Dates: First submitted 2025-02-06; First posted 2025-08-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Iron Absorption; Iron Requirements; Altitude
Keywords: iron absorption; altitude; stable iron isotopes; long-term iron balance

STUDY DESIGN:
Intervention Model Description: Two different groups of people residing at different altitudes will ingest the same amount of stable iron isotopes and during the observational period they will undergo the same measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isotopic labeled participants (Experimental): The two groups of participants differ only for their residence location at different altitudes. The intervention (administration of iron isotopes) does not differ among the two groups.
  Interventions: Dietary Supplement: Stable Isotopes

INTERVENTIONS:
Dietary Supplement: Stable Isotopes — 15 mg of stable iron isotopes in the form of ferrous sulphate 57FeSO4 will be orally administered to each participant.

SUMMARY:
Iron is an essential micronutrient responsible for a whealth of biological processes of the human body. Iron plays a fundamental role especially in oxygen transport, by binding to hemoglobin in the blood circulation. Iron intake from the diet needs to be in balance the unavoidable losses that occur daily via different pathways. The recommended daily requirement of iron is based on the balance between absorption and losses and is calculated to maintain a balance so that the absorption equals losses. At higher altitudes, the absorption of iron may be higher due to adaptation mechanisms in response to low oxygen concentration, and to maintain a larger erytroid compartement. However, the long-term effects of altitude on iron balance are unknown. Filling this knowledge gap is important to better understand iron deficiency in populations living at high and moderate altitudes. Therefore, the investigators plan to study people that live at two different altitudes and measure iron absorption and losses over the long term. This will be useful to formulate specific recommendations for this population groups, to expand the knowledge base to better prevent iron deficiency in Switzerland but also worldwide. Participants will be asked to consume a dose of stable iron isotopes. After one year from isotope administration, the isotopes will be equally distributed in all body compartments and any change in the isotope abundance with the normal occurring body iron can be detected. From this point onwards, the investigators can observe the iron turnover and calculate iron absorption and losses per unit of time. At 4 different visits blood samples will be taken from each participant.

DETAILED DESCRIPTION:
This study compares iron absorption in two population groups residing at different altitudes in Switzerland-one below 1000 meters above sea level and the other above 1500 meters. Additionally, the study aims to determine whether daily iron intake recommendations should be adjusted for high-altitude populations and to establish appropriate thresholds for diagnosing iron deficiency and iron deficiency anemia in these conditions. In each group 60 participants (30 men and 30 women) will be recruited. Each participant will be administered with an oral dose of iron isotopes in the form of ferrous sulphate 57FeSO4 dissolved in water. Ascorbic acid (vitamin C) will be additionally given with the isotope dose to increase the absorption and the enrichment in the body compartments and sirup will be added to the solution to confer a sweet flavour. There will be no other intervention throughout the course of the study.

The investigators will collect blood samples during the second year from study start at a frequency of 4 months for a total of 4 visits, at months 12, 16, 20 and 24. Venous blood samples for the measurement of the isotopic signal will be collected, and at two additional study visits the investigators will also measure hemoglobin using the so-called carbon monoxide (CO) rebreathing method that includes a CO rebreathing into a closed-circuit system in combination with pure oxygen. Before and after the 6 min re-breathing, capillary blood will be collected by finger prick in triplicates. At the study visits with blood withdrawal, the investigators will ask participants to fill questionnaires about dietary intake and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged 18-45 y
* BMI: 18 to 25 kg/m2
* Body weight <70 kg for females, <85 kg for males
* Plasma ferritin >25 µg/L
* Signed informed consent

Exclusion Criteria:

* Hb <12 g/dL (females), Hb <13 g/dL (males), corrected for altitude using the 2024 WHO guidance values for hemoglobin adjustments
* Inflammation (CRP > 5 mg/L)1
* Plasma ferritin >150 µg/L for females and >200 µg/L for males
* Chronic disease known to affect iron metabolism
* Chronic medications (except for oral contraceptives)
* Pregnancy (tested at screening) or intention to become pregnant during the course of the study
* Lactation
* High physical activity (MET-min/week > 3000 calculated according to the IPAQ, short version, administered at the screening)
* Difficulty with blood withdrawal
* Earlier participation in a study using stable iron isotopes or participation in any clinical study within the last 30 days
* Smoking
* Blood donation, blood transfusion or significant blood loss (more than 400 mL) over the past 6 months
* Intention to regularly donate blood during the 2 years duration of the study
* No residence in the respective location/altitude for at least the last 2 years
* No intention to reside in the respective location/altitude at least for the next 2 years
* Participants who are planning to spend an extended period (>12 weeks) at a different altitude from their residence location
* Spending more than 2 nights per week at a different location from residence location
* Inability to understand the information sheet and the informed consent form due to cognitive or language reasons

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
57Fe tracer concentration in the circulation | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  The measurement of the isotopic tracer concentration in the circulation allows to calculate the lon-term iron absorption in the participants, and the rate of change of the tracer allows to calculate the rate of change of body iron.

SECONDARY OUTCOMES:
Hemoglobin mass | 1 year after isotopic administration and every four months afterwards, for a total of 2 measurements for each participant.
  Hemoglobin mass will be measured using the CO-rebreathing method. In contrast to hemoglobin concentration, hemoglobin mass is more accurate since it does not depend on blood volume.
Ferritin concentration | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Ferritin concentration in serum, expressed as ug/L will be assessed as an indicator of the iron status.
Hepcidin concentration | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Hepcidin concentration in serum will be measured as a parameter for the iron status.
Serum transferrin receptor concentration | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  The serum concentration of the transferrin receptor (TfR) will be measure as a biomarker for iron status.
Concentration of c-reactive protein (CRP) | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Concentration of c-reactive protein (CRP) in mg/L will be measured in serum as a biomarker for inflammation status.
Concentration of alpha-1-acid glycoprotein (AGP) | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Concentration of serum AGP will be measured as abionarker for inflammation status
Concentration of erythropoietin | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Erythropoietin (EPO) concentration in whole blood will be measured as a biomarker for erythropoiesis.
Concentration of Erythroferrone (ERFE) | 1 year after isotopic administration and every four months afterwards, for a total of 4 measurements.
  Concentration of erythroferrone in serum will be measured as a biomarker for erythropoiesis.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, Prof. Dr., Principal Investigator — Fernfachhochschule Schweiz (FFHS), SUPSI
Locations (1):
- Fernfachhochschule Schweiz (FFHS), Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No